CLINICAL TRIAL: NCT06216535
Title: Escitalopram in Asthma Patients With Frequent Exacerbation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2023-0494; R61HL167909-01A1 (NIH)
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Escitalopram; SSRI; Adults
MeSH Terms: conditions — Asthma | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: This study is a two-arm, 26-week, randomized, single-center, double-blind, parallel group trial designed to evaluate the efficacy of treatment with escitalopram vs. placebo to reduce asthma exacerbations in n = 105 participants, ages 18-75 years, with moderate-to-severe asthma.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A randomization list will be maintained in a password-protected folder by an unblinded staff member with no participant contact and by the investigational pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive an inactive placebo by mouth using the same administration schedule as for escitalopram.
  Interventions: Drug: Placebo
- Escitalopram (Active Comparator): Participants will take oral escitalopram 10 mg per day for two weeks, followed by oral escitalopram 20 mg per day for 22 weeks. Participants will take oral escitalopram 10 mg per day for one week at the final study visit.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram is an FDA-approved SSRI antidepressant that is administered by mouth
  Arms: Escitalopram
Drug: Placebo — Inactive placebo comparator
  Arms: Placebo

SUMMARY:
Antidepressants, particularly selective serotonin reuptake inhibitors (SSRIs), such as escitalopram are widely used for mood and anxiety disorders. However, they have also been explored, with promising findings, for a variety of disorders outside of psychiatry. Clinical studies of SSRIs in depressed people with asthma were associated with decreased asthma exacerbations and improvement in asthma control. In this study, the number of asthma exacerbations will be assessed as the primary outcome measure in patients using escitalopram vs. placebo.

DETAILED DESCRIPTION:
A 26-week, randomized, double-blind, placebo-controlled trial of escitalopram will be conducted in 105 people with moderate to severe persistent asthma who, despite treatment with medium to high dose inhaled corticosteroids and long-acting beta-agonist therapy, had ≥ 3 asthma exacerbations in the past year. The primary outcome measure will be the number of times systemic corticosteroids are given for an asthma exacerbation with the Asthma Control Questionnaire as a secondary outcome measure. Mood and anxiety symptoms and functioning will be assessed as will the role of psychological asthma triggers on asthma symptom exacerbation. Serum IL-6 and peripheral eosinophil levels as well as fractional exhaled nitric oxide (FeNO) will be assessed. Thus, psychological/psychiatric and biological or immune mechanisms for the effect of escitalopram on asthma will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe persistent asthma
* Treatment with medium to high dose ICS and LABA therapy
* Three or more severe asthma exacerbations (requiring ≥ 3 days of systemic corticosteroids) in the past year
* Age 18-75 years old, male or female sex, English or Spanish speaking
* Participants will be required to be clinically stable with no recent exacerbations, infections or changes in asthma controller therapy for at least 4 weeks before study entry
* Biologic therapy for asthma (e.g., omalizumab, mepolizumab, reslizumab, benralizumab, dupilumab, tezepelumab) will be allowed if started at least 6 months prior to randomization

Exclusion Criteria:

* Current substance use disorder and/or current tobacco use or greater than 10 pack-years lifetime use
* A current MDD episode as well as bipolar disorder, schizophrenia, or schizoaffective disorder
* Vulnerable populations including intellectual disability or other severe cognitive impairment, inmates, pregnant or nursing women or women of childbearing age who will not use UT Southwestern IRB-approved methods of birth control or abstinence during the study
* Currently taking an antidepressant (antidepressants that are not SSRIs nor SNRIs prescribed for an indication other than depression at subtherapeutic doses are acceptable)
* High risk for suicide defined as > 1 past suicide attempts or any attempt within the past 12 months
* Severe or life-threatening medical illness that would make completion of study unlikely or clinically significant laboratory or ECG findings at baseline

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Total number of severe asthma exacerbations | 24 weeks
  A count outcome variable capturing the total number of severe asthma exacerbations. Severe asthma exacerbations will be defined by the use of oral corticosteroids ≥ 3 days, or hospitalization or emergency department visit leading to treatment with systemic glucocorticoids

SECONDARY OUTCOMES:
Asthma Control Questionnaire (ACQ) | 24 weeks
  The ACQ is a 7-item, self-report tool that measures asthma symptomatology over time. The ACQ assesses symptoms pertinent to the primary clinical goal of asthma management as identified by international guidelines including (a) day and nighttime symptoms, (b) activity limitation, (c) use of prn bronchodilators, and (d) FEV1% predicted.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D, Ph.D, MBA, Principal Investigator — UTSW Medical Center
Locations (1):
- UT Southwestern, 1440 Empire Central, Ste. LD4.100, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No